CLINICAL TRIAL: NCT02424461
Title: Antibiotic Treatment for 7 Days Versus 14 Days in Patients With Acute Male Urinary Tract Infection Due to Fluoroquinolones Susceptible Bacteria: a Multicentre, Non-inferiority, Double Blind, Randomized Placebo-controlled Trial
Brief Title: Antibiotic Treatment for 7 Days Versus 14 Days in Patients With Acute Male Urinary Tract Infection
Acronym: PROSTASHORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120116; AOM12268 (Other Grant/Funding Number: France: Ministry of Health (PHRC))
Record Dates: First submitted 2015-03-06; First posted 2015-04-23 (Estimated); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Acute Male Urinary Tract Infection
MeSH Terms: interventions — Ceftriaxone; Ofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 7 day-antimicrobial treatment (Active Comparator): Ceftriaxone : 1 injection 1 g per day for 2 days
  Ofloxacine : 400 mg/jour (200 mg/ jour in case of renal failure) for seven days
  Placebo of ofloxacine for 7 days
  Interventions: Drug: Ceftriaxone; Drug: Ofloxacine
- 14-day antimicrobial treatment (Active Comparator): Ceftriaxone : 1 injection 1 g per day for 2 days
  Ofloxacine : 400 mg/jour (200 mg/ jour in case of renal failure) for 14 days
  Interventions: Drug: Ceftriaxone; Drug: Ofloxacine; Drug: Placebo of ofloxacine

INTERVENTIONS:
Drug: Ceftriaxone — 1 injection 1 g per day for 2 days
Drug: Ofloxacine — 400 mg/jour (200 mg/ jour in case of renal failure) for seven days
Drug: Ofloxacine — 400 mg/jour (200 mg/ jour in case of renal failure) for 14 days
  Arms: 7 day-antimicrobial treatment
Drug: Placebo of ofloxacine — Placebo of ofloxacine for 7 days
  Arms: 14-day antimicrobial treatment

SUMMARY:
This study will investigate the treatment of urinary tract infection (UTI) in men. The investigators are looking to see if shorter duration of antibiotics (7 days) is not inferior to a longer duration of antibiotics (14 days). The investigators will also study whether longer treatment leads to an increase in antibiotic resistant bacteria in the gut microbiota or an increase in drug side effects.

DETAILED DESCRIPTION:
The proposed study is a multicentre, non-inferiority, double blind, randomized placebo-controlled trial of treatment duration for male urinary tract infection (UTI) due to fluoroquinolones susceptible bacteria. Specifically, 284 men with a UTI will be randomized to 7 vs. 14 days of antimicrobial treatment. The primary outcome is resolution of fever, sterile urine analysis 4 weeks after completion of antimicrobial therapy and no antibiotic therapy active against the bacterial strain responsible for the UTI within the 4 week period following antimicrobial therapy. Secondary outcomes include the intestinal carriage of antimicrobial-resistant Gram-negative bacilli at the end of treatment, the incidence and severity of adverse drug events and the recurrent UTI within the treatment period and 4 weeks and 12 weeks of completing active study medication.

Currently, the optimal treatment duration for male UTI is unknown. Only one randomized study showed no difference in outcomes, in patients treated with ciprofloxacin during 14 vs. 28 days. However, this study was underpowered and included patient in a single center. Current treatment guidelines are not consensual and recommend treating men with UTI for 7 to 4 or 6 weeks. Shorter durations may expose patients to recurrence when longer duration may be associated with increase in Clostridium difficile infection and antimicrobial resistance. Longer-duration treatment is also more costly and inconvenient to patients. Thus, since longer-duration treatment is associated with some adverse outcomes, in order to justify longer-duration treatment thee must be some clinically significant benefit to the extended treatment.

The proposed randomized placebo-controlled trial will test the hypothesis that 7 days of antimicrobial treatment is non-inferior for the resolution of fever and microbiological success when compared to 14 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male gender, 18 years and older
* New-onset of the following criteria:

  1. Temperature ≥38° Celsius or <36° Celsius (or at least once in the 3 previous days), AND
  2. at least one of following symptoms/findings: dysuria, urinary frequency, urgency, urinary burning, hematuria, perineal pain, supra-pubic pain or urinary retention, painful prostate (digital prostate examination)
* Leucocyturia ≥ 10/ mm3
* Urinary signs/symptoms within the 3 previous months
* Urinary culture yielding a single pathogen, at least10^3 colony-forming unit (CFU)/ml, susceptible to nalidixic acid, ofloxacine and ceftriaxone.
* Oral route for study drug
* Normal Ultrasound prostatic findings (no abscess and post-void residual urine volume < 100 ml).

Exclusion Criteria:

* Septic shock
* Admission to the hospital (for > 48 h) at the time of diagnosis
* Treatment for UTI in the past year
* Urinary catheter
* Severe disease with strong probability of death within 3 months
* Severe allergy or contraindication to fluoroquinolones or beta-lactams
* Not able to give informed consent
* Antimicrobial therapy with fluoroquinolone or aminoglycoside in the 3 previous days
* Neutropenia (neutrophils count < 500/mm3)
* Renal insufficiency (creatinin clearance ≤ 20 ml/min)
* Glucose - 6 - Phosphate - Dehydrogenase deficiency
* Significant cognitive disorders
* Uncontrolled epilepsy
* History of tendinitis
* Elevated liver enzyme levels (aspartate aminotransferase (ASAT), Alanine Amino Transferase (ALAT) ≥ 5 upper limit of normal range (ULN))
* Myasthenia
* Significant psychiatric disorders
* Galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.
* Patient under guardianship patient, guardianship or without social security cover

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2015-01-25 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
Success defined by resolution of fever | day 42
  Defined by 3 criteria that should be fulfilled:
  1. resolution of fever between the end of treatment and 4 weeks thereafter (except fever not related to urine infection),
  2. sterile urine (except alpha-hemolytic streptococus, Lactobacillus, Corynebacterium, Gardnerella or coagulase negative Staphylococcus) analysis 4 weeks after completion of antimicrobial therapy, and
  3. no antibiotic therapy active against the bacterial strain responsible for the UTI within the 4 week period following antimicrobial therapy

SECONDARY OUTCOMES:
Intestinal carriage of antimicrobial-resistant Gram-negative bacilli | 4 and 12 weeks
  intestinal carriage of antimicrobial-resistant Gram-negative bacilli at the end of treatment and 4 and 12 weeks after completing study medication, as compared to a baseline sample taken before treatment
Incidence and severity of adverse drug events | 4 and 12 weeks
  the incidence and severity of adverse drug events within the treatment period and in the 4 and 12 weeks after completing study medication
Recurrent UTI | 4 and 12 weeks
  Recurrent UTI within 4 weeks and 12 weeks of completing active study medication

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis hospital, Paris, France

REFERENCES:
- [Background] Lafaurie M, Chevret S, Fontaine JP, Mongiat-Artus P, de Lastours V, Escaut L, Jaureguiberry S, Bernard L, Bruyere F, Gatey C, Abgrall S, Ferreyra M, Aumaitre H, Aparicio C, Garrait V, Meyssonnier V, Bourgarit-Durand A, Chabrol A, Piet E, Talarmin JP, Morrier M, Canoui E, Charlier C, Etienne M, Pacanowski J, Grall N, Desseaux K, Empana-Barat F, Madeleine I, Bercot B, Molina JM, Lefort A; PROSTASHORT Study Group. Antimicrobial for 7 or 14 Days for Febrile Urinary Tract Infection in Men: A Multicenter Noninferiority Double-Blind, Placebo-Controlled, Randomized Clinical Trial. Clin Infect Dis. 2023 Jun 16;76(12):2154-2162. doi: 10.1093/cid/ciad070. PMID 36785526